CLINICAL TRIAL: NCT06066931
Title: Reconstruction of the Pelvic Floor and Perineal Wound After Extralevatory Abdominal-perineal Extirpation of the Rectum
Brief Title: Reconstruction of the Pelvic Floor and Perineal Wound After Rectal ELAPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuban State Medical University (Other)
Collaborators: State Budget Public Health Institution Scientific Research Institute - Ochapovsky Regional Clinical Hospital (Other Government); City Clinical Oncology Hospital No 1 (Other Government)
Responsible Party: Principal Investigator, Vadim Polovinkin, Doctor of Medical Sciences, Head of the Department of General Surgery of Kuban State Medical University, Kuban State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28092023
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Rectum Cancer
Keywords: Cancer of the lower ampullary rectum; Extralevatory abdominal-perineal extirpation; Plastic surgery of the pelvic floor and perineal wound
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: It is planned to recruit patients over the age of 18, suffering from cancer of the lower ampullary rectum with T1-T4N0-2M0 (according to the classification of malignant tumors TNM in the 8th edition) who meet the inclusion criteria taking into account the exclusion criteria in the number of 150 people. Group 1 is a simple method (Plastic surgery with local tissues) n=50; Group 2 is plastic surgery with a mesh endoprosthesis n=50; group 3 is a new method of plastic surgery n=50.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 of a simple method (Plastic surgery with local tissues) n=50 (Other): In group 1 patients (plastic surgery with local tissues), a simple layer-by-layer suturing of the sciatic-anal and subcutaneous adipose tissue is performed using nodular sutures. The skin was sewn up with nodular sutures at the discretion of surgeons. The installation of abdominal drainage and/or perineal drainage was left to the discretion of the surgeon.
  Interventions: Procedure: Plastic surgery of the pelvic floor and perineal wound with local tissues
- Group 2 is plastic surgery with a mesh endoprosthesis n=50 (Other): In group 2 patients, a mesh allograft with an adhesive coating is inserted into the bottom of the wound, positioned horizontally between the inner surfaces of the ischial bones and vertically between the sacrum and the vagina in women or between the sacrum and the prostate gland in men. The mesh was sewn from behind on both sides of the coccyx or sacrum. From the side, the mesh was attached to the remainder of the levator muscle and from the front to the transverse muscles of the perineum. The installation of abdominal drainage and/or perineal drainage was left to the discretion of the surgeon. The sciatic-anal and subcutaneous fat are sutured using nodular sutures.
  Interventions: Procedure: Plastic surgery of the pelvic floor and perineal wound with mesh endoprosthesis
- Group 3 is a new method of plastic surgery n=50 (Experimental): In group 3 the plastic stage is performed: on one side of the perineal wound, a cutaneous-subcutaneous-fascial flap on the leg is cut out and deepithelized, along the entire length of the wound, thereby forming a diamond-shaped perineal wound, plunging it into the pelvic aperture, fixing it with single sutures to the remnants of the muscle lifting the anus of the opposite side, and the flap width is 3-4 cm to fill the pelvic aperture. On the opposite side of the wound, a triangular skin-subcutaneous fascial flap is cut out on a leg equal to the width of the previously formed diamond-shaped wound at an angle of 60-80 degrees from the middle of the wound edge, and the sides of the triangular flap should be equal to half the length of the edge of the diamond-shaped wound, then it is moved and additionally fill the wound cavity with it, in condition of displacement of the apex of the triangle flap with the top of the rhombus-wounds. The flap is fixed with separate skin nodular sutures.
  Interventions: Procedure: Plastic surgery of the pelvic floor and perineal wound with counter-displaced skin-subcutaneous fascial flaps after extralevatory abdominal-perineal extirpation of the rectum

INTERVENTIONS:
Procedure: Plastic surgery of the pelvic floor and perineal wound with counter-displaced skin-subcutaneous fascial flaps after extralevatory abdominal-perineal extirpation of the rectum — Skin-subcutaneous fascial flap on the leg is cut out from one side of the perineal wound, and deepithelized, forming a diamond-shaped perineal wound. The cut flap is immersed in the aperture of the pelvis and fixed with single sutures to the remains of levators of the opposite side. The flap width should be 3-4 cm, sufficient to fill the pelvic aperture. On the opposite side of the wound, a skin-subcutaneous fascial flap is cut out on a triangular leg equal to the width of the previously formed diamond-shaped wound. The flap is moved to the center of the wound, additionally filling wound cavity with it, combining the vertex of the triangle with the vertex of the rhombus. The perineal wound is drained through the contraperture. The flap is fixed with separate nodal seams.
  Arms: Group 3 is a new method of plastic surgery n=50
Procedure: Plastic surgery of the pelvic floor and perineal wound with local tissues — Simple layer-by-layer suturing of the sciatic-anal and subcutaneous adipose tissue is performed using nodular sutures. The skin was sewn up with nodular sutures at the discretion of surgeons. The installation of abdominal drainage and/or perineal drainage was left to the discretion of the surgeon.
  Arms: Group 1 of a simple method (Plastic surgery with local tissues) n=50
Procedure: Plastic surgery of the pelvic floor and perineal wound with mesh endoprosthesis — A mesh allograft with an adhesive coating is inserted into the bottom of the wound, positioned horizontally between the inner surfaces of the ischial bones and vertically between the sacrum and the vagina in women or between the sacrum and the prostate gland in men. The mesh was sewn from behind on both sides of the coccyx or sacrum. From the side, the mesh was attached to the remainder of the levator muscle and from the front to the transverse muscles of the perineum. The installation of abdominal drainage and/or perineal drainage was left to the discretion of the surgeon. The sciatic-anal and subcutaneous fat are sutured using nodular sutures.
  Arms: Group 2 is plastic surgery with a mesh endoprosthesis n=50

SUMMARY:
A multicenter, cohort, randomized, controlled study is being conducted since the 1of September, 2023 whereby the immediate and long-term results of pelvic floor and perineal wound plastic surgery after extralevatory abdominal-perineal extirpation of the rectum will be compared. The study is conducted on the basis of the Federal State Budgetary Educational Institution of the Ministry of Health Care of the Russian Federation, the Department of General Surgery at the clinical base of the State Budgetary Healthcare Institution " Krasnodar Regional Hospital No. 1 named after Professor S.V. Ochapovsky" of the Ministry of Health Care of the Krasnodar Territory, State Budgetary Healthcare Institution " Krasnodar Oncological Dispensary No. 1" of the Ministry of Health Care of the Krasnodar Territory The study included patients over 18 years old suffering from cancer of the lower ampullary rectum with T1-T4N0-2M0 (according to the classification of malignant tumors TNM in the 8th edition), who are scheduled for extralevatory abdominal-perineal extirpation of the rectum. Patients are randomized into 3 groups: the first group includes patients with plastic surgery in a simple way (Plastic surgery with local tissues), the second group includes patients with plastic surgery with a mesh endoprosthesis and the third one includes patients with plastic surgery in a new way.

The purpose of the study is to evaluate the effectiveness of the developed method of pelvic floor and perineal wound plastic surgery after extralevatory abdominal-perineal extirpation of the rectum. It is easily reproducible and provides high-quality closure of the deep and skin defect of the perineal wound. In addition, the new method will reduce the frequency of postoperative complications when compared with the use of conventional methods of closing the defect of the perineum, the method improves the quality of life and provides early rehabilitation of patients.

Study status- patients are being recruited. Number of patients selected is 150 patients. The primary endpoint of the study is the assessment of the early postoperative period and the frequency of postoperative complications (Flap necrosis; Suppuration; Hematoma; Bleeding; Seroma) within 30 days from the date of surgery. The study was approved by the Independent Ethics Committee Protocol No. 112 of 12th November, 2022.

It is planned to recruit patients within 2 years and monitor each of them for 30 days after surgery to assess the primary endpoint and to monitor patients within 1 year to assess the secondary endpoint. The secondary endpoint means an assessment of the frequency of late postoperative complications (perineal fistula, abscess, hernia) and an assessment of the quality of life within 1 year after surgery. It is planned to complete the study in 2025.

Eventually it is planned to publish the protocol of the study, the results obtained after the recruitment of the required number of patients as well as the results of evaluation of the primary endpoint.

DETAILED DESCRIPTION:
The aim of the study is to improve the results of pelvic floor and perineal wound plastic surgery after extralevatory abdominal-perineal extirpation (EAPE) of the rectum for cancer of the lower ampullary rectum by applying a new method of plastic surgery.

Being examined according to the standards of cancer treatment of the lower ampullary part of rectum, patients are hospitalized in the oncological surgery department. In the preoperative period, they are randomized by the Randomizer program into 3 groups by the head of the study on the day of surgery: the 1st Group includes patients to be made plastic surgery in a simple way (Plastic surgery with local tissues), the 2nd Group includes patients to be made plastic surgery with a mesh endoprosthesis and the 3rd Group includes patients to be made plastic surgery in a new way.

Patient data, clinical trial results, and randomization results are introduced into the Microsoft Access database.

The operation is carried out as follows: under combined endotracheal anesthesia after the completion of the abdominal and pelvic stage of the operation ending with the mobilization of the rectum which is carried out along the posterior wall to the level of V sacral vertebra corresponding to the bend of the sacrum; along the anterior wall that is the level of seminal vesicles, the upper pole of the prostate gland in men, the middle third of the vagina in women; along the lateral walls reaching the level of the pelvic nerve plexus and finally a single-stem colostomy is formed.

Suturing of the wound of the anterior abdominal wall with drainage of the pelvic cavity is performed. The patient is placed on his abdomen with his legs apart - "the position of a penknife". The operating surgeon is positioned between the patient's legs. Suturing of the skin of the perianal area with a pouch suture is performed after surgical treatment and limitation of the surgical area. Re-processing of the operating area is performed. It is made a fringing incision in the perianal region from the level of the sacrococcygeal joint, along the perianal-skin folds to the middle of the perineal seam. 2-4 sutures of wound fiber fixing to the skin of the external gluteal region may be applied for the purpose of additional traction in patients with severe obesity.

Cylindrical mobilization of the rectum is performed with the capture of sciatic-rectal fiber and the external sphincter along the posterior and lateral walls. If necessary, to improve visualization or in case of tumor invasion, the coccyx is amputated. After crossing the sacro-rectal and anococcygeal ligaments, they are connected to the abdominal cavity. The pelvic tendon arch is sequentially crossed along the posterolateral walls, with a transition to the side walls and a wide cut-off of the muscle that raises the anus from the fixation site to the sciatic bone. After mobilization of the posterior and lateral semicircles, the drug is turned into the perineal wound and mobilization is continued along the anterior semicircle. After removal of the rectum with a neoplasm, the part of it is sent for histological examination. The cavity of the perineal wound is sanitized with an antiseptic solution. The plastic stage of the operation is performed: - In group 1 patients (plastic surgery with local tissues), a simple layer-by-layer suturing of the sciatic-anal and subcutaneous adipose tissue is performed using nodular sutures. The skin was sewn up with nodular sutures at the discretion of surgeons. The installation of abdominal drainage and/or perineal drainage was left to the discretion of the surgeon.

- In group 2 patients, a mesh allograft with an adhesive coating is inserted into the bottom of the wound, positioned horizontally between the inner surfaces of the ischial bones and vertically between the sacrum and the vagina in women or between the sacrum and the prostate gland in men. The mesh was sewn from behind on both sides of the coccyx or sacrum. From the side, the mesh was attached to the remainder of the levator muscle and from the front to the transverse muscles of the perineum. The installation of abdominal drainage and/or perineal drainage was left to the discretion of the surgeon. The sciatic-anal and subcutaneous fat are sutured using nodular sutures.

In group 3 patients, the plastic stage is performed as follows: on one side of the perineal wound, a cutaneous-subcutaneous-fascial flap on the leg is cut out and deepithelized, along the entire length of the wound, thereby forming a diamond-shaped perineal wound, plunging it into the pelvic aperture, fixing it with single sutures to the remnants of the muscle lifting the anus of the opposite side, and the flap width is 3-4 cm, sufficient to fill the pelvic aperture. On the opposite side of the wound, a triangular skin-subcutaneous fascial flap is cut out on a leg equal to the width of the previously formed diamond-shaped wound at an angle of 60-80 degrees from the middle of the wound edge, and the sides of the triangular flap should be equal to half the length of the edge of the diamond-shaped wound, then it is moved and additionally fill the wound cavity with it, in condition of displacement of the apex of the triangle flap with the top of the rhombus-wounds. The perineal wound is drained through the contraperture. The flap and the edges of the wound are separated from the gluteal muscles and the flap is fixed with separate skin nodular sutures to eliminate tension.

The results of the operation, the postoperative course and the quality of life are recorded in the Microsoft Access database with subsequent statistical processing. The postoperative wound photo is made in the day of discharge (up to 30 days after surgery).

Expected results: after completing the recruitment of patients to the comparison groups and after statistical processing it is planned to obtain an evidence base on reducing the frequency of early and late postoperative complications in the group with plastic surgery in a new way.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old suffering from cancer of the lower ampullary rectum cT1-T4N0-2M0 (according to the classification of malignant tumors TNM in the 8th edition).
2. Patients with planned extralevatory abdominal-perineal extirpation of the rectum.
3. Physical status of patients according to ASA classification I-II.
4. Signed informed consent to participate in the study.

Non-inclusion criteria:

1. Verification of the squamous cell carcinoma diagnosis.
2. The presence of acute purulent processes in the area of surgical intervention.

Exclusion Criteria:

1. Refusal to participate at any stage of the study.
2. Death in the early postoperative period (up to 30 days after surgery) caused by somatic complications not associated with surgery (PATE, myocardial infarction, stroke).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The assessment of the frequency of early postoperative complications | Within 30 days from the date of surgery
  Early postoperative complications to be assessed: flap necrosis; suppuration; hematoma; bleeding; seroma

SECONDARY OUTCOMES:
The assessment of the frequency of late postoperative complications and quality of life | Within 1 year after surgery
  Late postoperative complications to be assessed: perineal fistulas, abscesses, hernias

CONTACTS AND LOCATIONS:
Overall Officials: Vadim V Polovinkin, MD, Principal Investigator — Kuban State Medical University

IPD SHARING:
Plan to Share IPD: No
An IPD sharing plan will be determined after start of the clinical trial.